CLINICAL TRIAL: NCT01071148
Title: A Phase IV, Prospective, Observational, Open Label, Single Centre Cohort Trial to be Conducted in Norway During One Year to Assess the Cumulative Pregnancy Rate in a New Series of In-vitro Fertilization (IVF) Treatment Cycles Following Three or More Previous IVF Treatment Cycles Without Live Birth.
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Norway (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR200061-502; 2008-002840-41 (EudraCT Number); NCT00893204 (obsolete NCT alias)
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Infertility
Keywords: Infertility; Gonal-f; Pergoveris; Luveris
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subgroup 1: Age < 35 years: Subjects who have experienced infertility and justifying IVF/ET treatment will be administered either Gonal-f or Pergoveris or Gonal-f and Luveris as per the discretion of the investigator.
- Subgroup 2: 42 > Age ≥ 35 years: Subjects who have experienced infertility and justifying IVF/ET treatment will be administered either Gonal-f or Pergoveris or Gonal-f and Luveris as per the discretion of the investigator.

SUMMARY:
The primary objective of this observational study is to assess the cumulative rate of ongoing pregnancy at 10 ±2 weeks after hCG administration in a new series of IVF-treatment cycles in a total of 176 subjects, who have undergone three or more previous IVF-treatment cycles without live birth. Secondary objectives include subgroup analysis on the effect of age on the likelihood of pregnancy at 10 ±2 weeks after hCG administration in a new series of IVF-treatment cycles in patients < 35 years and ≥ 35 years, who have undergone three or more previous IVF-treatment cycles without live birth.

The information obtained from this trial will be helpful for subjects who are considering further IVF treatments and for IVF centres, as well as for the formulation of governmental policies regarding healthcare reimbursement in Norway.

DETAILED DESCRIPTION:
Since IVF processes were established in 1978, there has been a dramatic increase in the numbers of IVF treatment cycles performed worldwide. In 2003, the total numbers of reported IVF cycles were 132,932 from 725 clinics in 28 European countries, 7,535 IVF/intra cytoplasmic sperm injection (ICSI) cycles from 24 centres in Canada, and over 100,000 IVF cycles from 399 centres in the U.S.

Of all the assisted reproductive technology (ART) procedures available, IVF leads to the highest pregnancy rate per cycle. The degree to which governments reimburse subjects for IVF treatment varies widely among countries in Europe and North America. In Norway, infertile subjects are offered a maximum of three IVF-cycles reimbursed by the government. If three cycles are unsuccessful, subjects must pay for further treatments. This policy might lead subjects to believe that the probability of achieving pregnancy after four or more cycles is very low and, therefore, not worth the cost or effort.

However, a number of published studies show evidence of successful outcomes for additional IVF-cycles after three (or more) cycles with negative results. Many studies show only a modest decline of success with repeated IVF cycles. In addition, a preliminary retrospective analysis of the clinical pregnancy rate in subjects treated at the trial centre during 2007 showed that subjects, who underwent additional one to three IVF-treatment cycles, had a cumulative success rate of 52% (based on clinical experience from 62 subjects at the Hausken clinic in 2007). Thus, these studies indicate that there is a reasonable chance of achieving a healthy pregnancy and live birth after three previous IVF-treatment failures.

In fact, age is likely to be a more important factor than the number of previous IVF treatment failures in determining a successful outcome. Several studies have demonstrated that older women have lower rates of conception and live births, and higher rates of pregnancy failure.

Treatment of subfertility and infertility by ART such as IVF and embryo transfer (ET) requires multiple follicular development to increase the number of female gametes, and the chances of a successful treatment outcome. Ovarian stimulation in IVF/ICSI currently includes suppression of endogenous luteinising hormone (LH) secretion by administration of a gonadotropin releasing hormone (GnRH) analogue, followed by stimulation of multiple follicular development by exogenous follicular stimulating hormone (FSH) administration. When adequate follicular development is achieved, a single dose of human chorionic gonadotropin (hCG) or LH is administered to mimic the endogenous LH surge and induce oocyte maturation.

A total of 176 subjects who had previously undergone three or more IVF-treatment cycles that did not result in live birth will undergo a new series of IVF-treatment cycles using Gonal-f or Pergoveris or Gonal-f and Luveris. Subjects both < 35 years and ≥ 35 years will be included. Subgroup analysis will take into account the effect of age on the likelihood of success after repeated cycles of IVF. The investigators will systematically follow-up these subjects to observe their cumulative ongoing pregnancy rate.

The study will consist of a screening period (≤-4months) during which the following trial assessments will be made: demographics, medical history, concomitant medications, clinical examination, vital signs, number of antral follicles and a subject diary will be handed out to the subjects. Between screening and the beginning of treatment, there will an optional telephone consultation during which any screening information or changes in concomitant medications will be updated. Down-regulation treatment will start within 3 months following the screening visit during the pre treatment period with GnRH daily agonist or antagonist commercially available in Norway, for pituitary gonadotrope cell desensitisation. FSH treatment will begin by administering either Gonal-f or Pergoveris or Gonal-f and Luveris after at least 2 weeks of GnRH agonist down-regulation. If a GnRH antagonist protocol is used, FSH injections will start on Day 2 of the menstrual cycle.

Follicular development will be monitored according to the centre's standard practice by ultrasound and/or estradiol (E2) levels, until the protocol hCG requirement is met (i.e. at least 1 follicle ≥18 mm and 2 follicles ≥16 mm) at which time the subject will receive hCG (Day 0), according to the routine practice of the centre, in order to induce final oocyte maturation. Ovum Pick Up (Day 2), IVF, ET (Day 4-7) and luteal phase support will be performed as per the centre's standard practice. During the treatment period several assessments will be made and any adverse events (AEs) observed during the trial will be recorded. A urine pregnancy test will be performed 16 days post hCG administration. In case of negative urine pregnancy test, the subject will be assessed for the post-treatment safety follow-up and the cycle will be considered as 'completed'. The post-treatment safety follow-up can take place simultaneously with the next cycle's screenings visit. If subject drops out, the early termination visit will replace the post-treatment safety follow-up. If the urine pregnancy test is positive, clinical and later ongoing pregnancy will be subsequently confirmed by ultrasound scan according to the centre's routine practice. At this last visit, all subjects will be assessed for the post-treatment safety follow-up and will be considered 'completed'. Pregnancy outcome in pregnant subjects will be optionally followed up until delivery.

Adverse events and serious adverse events (SAEs) will be assessed if spontaneously reported by the subjects at all study visits: during an optional telephone consultation between screening and the beginning of treatment, ultrasound scan (Day -7-0), OPU (Day 2), telephone consultation (Day 3), embryo transfer (Day 4-7), telephone consultation (Day 16), scan week 12 (assessed 10 weeks after hCG administration), post-treatment safety follow-up, 1-Year follow-up, and at early termination (if applicable).

ELIGIBILITY:
Inclusion Criteria:

* Infertility justifying IVF/ET treatment
* The decision of treating subject with GONAL-f or Pergoveris or GONAL-f and Luveris is made before considering the subject for the trial.
* Age between 18th and 42nd birthday at the screening visit.
* Have undergone three or more previous IVF-treatment cycles that did not result in live birth.
* Have good general health that allows IVF therapy
* Have a male partner with semen analysis, performed within 12 months prior to screening, that was considered adequate to proceed with regular insemination or ICSI according to the centre's standard practice
* At least one ovary present
* Have given written informed consent

Exclusion Criteria:

* FSH > 12 IU/L
* Body mass index (BMI) > 40 kg/m2
* Pre-treatment antral follicle count [follicles ≥2mm - <11mm]) < 4
* Previous IVF attempts with no follicle development.
* Any contraindication for the use of GONAL-f or Pergoveris or Luveris (refer to SPC)

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total of 176 subjects justifying IVF therapy at a single IVF centre in Norway will be recruited into this trial. Subjects must have been treated with three or more previous IVF-cycles without live birth.
Sampling Method: Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2009-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Cumulative ongoing pregnancy rate within one year of starting the trial in the total trial population | 10 ± 2 weeks after hCG administration
  Ongoing pregnancy is defined as the existence of at least one ultra-sonographically-confirmed gestational sac in the uterus, with foetal heart activity

SECONDARY OUTCOMES:
Number of mature follicles of ≥18 mm in size | 7 days before hCG administration till the day of hCG administration i.e.day (-)7 - 0
Number of oocytes retrieved | Day 2
Fertilisation rate | Day 3
Positive pregnancy test per cycle and cumulatively | 16 days post hCG administration
Cumulative clinical pregnancy rate within one year of starting the trial | 5 weeks ± 2 weeks after hCG administration
Clinical pregnancy rate per first, second and third new IVF-cycle | 5 weeks ± 2 weeks after hCG administration
Ongoing pregnancy rate per first, second and third new IVF-cycle | 10 weeks ± 2 weeks after hCG administration
Cumulative live birth rate(if available) | Follow-up period of 1 year
Cumulative ongoing pregnancy rate within one year of starting the trial in subjects aged < 35 years and ≥ 35 years | 10 ± 2 weeks after hCG administration
  Ongoing pregnancy is defined as the existence of at least one ultra-sonographically-confirmed gestational sac in the uterus, with foetal heart activity
Ongoing pregnancy rate per IVF-treatment cycle within one year of starting the trial in the total trial population and in subgroup analysis in subjects aged < 35 years and ≥ 35 years | 10 ±2 weeks after hCG administration

CONTACTS AND LOCATIONS:
Overall Officials: Viveka Åberg, MD, Study Director — Merck Serono Norway
Locations (1):
- Klinikk Hausken, Haugesund, Norway